CLINICAL TRIAL: NCT02700516
Title: Recurrent Primary Glomerulonephritis After Renal Transplantation: Effects on Renal Allografts and Transplant Recipients
Brief Title: Recurrent Glomerulonephritis After Renal Transplantation
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Caliskan, Associate Professor of Medicine, Istanbul University
Other Study IDs: 32364/200
Record Dates: First submitted 2016-02-25; First posted 2016-03-07 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Recurrent GN: Renal transplant recipients with biopsy-confirmed recurrent primary glomerulonephritis.
- Non-recurrent GN: Renal transplant recipients with non-recurrent primary glomerulonephritis.
- Non-GN: Renal transplant recipients with etiologies other than primary glomerulonephritis.

SUMMARY:
Glomerulonephritis (GN) is the leading cause of end-stage renal disease in 30% to 50% of patients who receive a renal transplant. The exact prevalence of either recurrent or de novo GN is unknown since a considerable number of patients never undergo allograft biopsy, leaving GN underdiagnosed. The aim of this study is to evaluate the effects of recurrent GN on the prevalence, risk factors, clinicopathological features, and outcome of renal transplant recipients.

DETAILED DESCRIPTION:
Glomerulonephritis is the leading cause of end-stage renal disease in 30% to 50% of patients who receive a renal transplant. Even though recurrent or de novo posttransplant primary GN is the third most frequent cause of renal allograft loss after renal transplantation, different recurrence rates have been reported in different patient series worldwide. With the implementation of diverse and improved immunosuppressive treatment regimens and prolongation of graft survival, renal allograft loss caused by recurrent or de novo GN will be more important than ever. Data obtained from comparing patients who have recurrent primary GN against patients with non-recurrent GN and renal transplant recipients with non-GN etiology shall bring new approaches to the daily practice of managing patients with GN and renal failure, assessing them as transplant candidates and applying new therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a renal transplantation because of an end-stage renal disease caused by primary glomerulonephritis and have biopsy-proven recurrent primary glomerulonephritis (Recurrent GN group)
* Patients who underwent a renal transplantation because of an end-stage renal disease caused by primary glomerulonephritis and have no signs of recurrence (Non-recurrent GN group)
* Patients who underwent a renal transplantation because of an end-stage renal disease linked to an etiology other than primary glomerulonephritis (Non-GN group)

Exclusion Criteria:

* Patients who are unwilling or unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Allograft survival | 1 - 5 years

SECONDARY OUTCOMES:
Allograft rejection | 1 - 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Caliskan, MD, Principal Investigator — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul
  - Division of Nephrology, Department of Internal Medicine, Cerrahpasa Faculty of Medicine, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Briganti EM, Russ GR, McNeil JJ, Atkins RC, Chadban SJ. Risk of renal allograft loss from recurrent glomerulonephritis. N Engl J Med. 2002 Jul 11;347(2):103-9. doi: 10.1056/NEJMoa013036. PMID 12110738